CLINICAL TRIAL: NCT00165867
Title: An Open Label Phase II Study of Indisulam in Combination With Irinotecan in Patients With Metastatic Colorectal Cancer Who Have Been Previously Treated With 5-Fluorouracil/Leucovorin and Oxaliplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7070-E044-214
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2006-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — N-(3-chloro-7-indolyl)-1,4-benzenedisulphonamide

INTERVENTIONS:
Drug: E7070

SUMMARY:
The overall purpose of this study is to determine the efficacy, safety and tolerability of indisulam in combination with irinotecan as a treatment for patients with metastatic colorectalcancer previously treated with 5-fluorouracil/leucovorin and oxaliplatin (FOLFOX).

ELIGIBILITY:
Inclusion criteria:

* Ambulant male or female patients with metastatic colorectal cancer who have been previously treated with 5-fluorouracil/leucovorin and oxaliplatin. Patients must fulfill the following criteria to be included in the study:
* At least 4 doses of previous treatment with oxaliplatin
* All previous treatment (including surgery and radiotherapy) must have been completed at least four weeks prior to study entry and any acute toxicities must have resolved
* At least one uni-dimensionally measurable lesion according to RECIST criteria (the following do not qualify as measurable lesions: bone, leptomeningeal disease, ascites, pleural/pericardial effusion, lymphangitis cutis/pulmonis, abdominal masses that are not confirmed and followed by imaging techniques, and cystic lesions)
* Aged greater than or equal to 18 years
* Histologically or cytologically confirmed colorectal cancer
* Karnofsky performance status greater than or equal to 70%
* Written informed consent to participate in the study

Exclusion criteria:

Patients with the following characteristics will not be included in the study:

* More than three previous lines of chemotherapy (including neo-adjuvant and adjuvant)
* Prior treatment with cytotoxics other than 5- fluorouracil/leucovorin (capecitabine and UFT are permitted) and oxaliplatin. Prior epidermal growth factor receptor targeted and anti-angiogenic therapy is permitted.
* Untreated brain metastases (patients who have been treated for CNS metastases must be asymptomatic and radiologically stable for 4 weeks prior to entry). Patients must not have clinical symptoms from brain metastases and must not be taking corticosteroids for the treatment of brain metastases. Patients must not have leptomeningeal metastases
* Any of the following laboratory parameters:

  1. hemoglobin <10 g/dl;
  2. neutrophils <1.5 x 109/L;
  3. platelets <100 x 109/L;
  4. serum bilirubin >25 mmol/l (1.5 mg/dl);
  5. other liver parameters >2.5 x upper normal limit (ULN) (> 5 x upper normal limit in the presence of hepatic metastases);
  6. serum creatinine >1.5 x ULN;
  7. serum calcium (corrected for albumin) >=11.5 mg/dl. 5. History of Gilbert's Disease or conjugated hyperbilirubinemia 6. Concurrent or previous malignancy of a different tumor type within five years of starting the study except for adequately treated non- melanoma skin cancer or cervical intraepithelial neoplasia
* Uncontrolled infections
* Clinically significant cardiac impairment or unstable ischemic heart disease including a myocardial infarction within six months of study start
* Chronic inflammatory bowel disease and/or bowel obstruction
* History of hypersensitivity to sulfonamides
* History of severe hypersensitivity reactions to one of the excipients of irinotecan
* Treatment within two weeks before the start of the stud y with any of the following: coumarin anti-coagulants, terfenadine, cisapride, cyclosporin, tacrolimus, theophylline, diazepam, sulphonylurea hypoglycaemics, phenytoin, or carbamazepine
* Any treatment with investigational drugs within 30 days before the start of the study
* Pregnancy or lactation (all women of childbearing potential must have a negative pregnancy test before inclusion in the study; post-menopausal women must be amenorrheic for at least 12 months). Female patients must use adequate contraceptive protection
* Fertile males not willing to use contraception or whose female partners are not using adequate contraceptive protection
* History of alcoholism, drug addiction, or any psychiatric or psychological condition which, in the opinion of the investigator, would impair study compliance.
* Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-04

PRIMARY OUTCOMES:
The objective response rate as defined by RECIST criteria.

SECONDARY OUTCOMES:
Duration of response
time to progression
overall survival
safety and tolerability of the combination

CONTACTS AND LOCATIONS:
Overall Officials: Jantien Wanders, Study Director — Eisai Limited
Locations (7):
- France (3):
  - Hôpitaux Civils de Colmar, Colmar
  - CRLC Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
- United Kingdom (4):
  - Aberdeen Royal Infirmary, Aberdeen
  - Beatson Oncology Centre, Glasgow
  - Cookridge Hospital, Leeds
  - Leicester Royal Infirmary, Leicester